CLINICAL TRIAL: NCT04396119
Title: Developing Lung Cancer Screening in Hodgkin Lymphoma Survivors: a Qualitative Study
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp178; 276443 (Other: IRAS Project ID)
Record Dates: First submitted 2020-01-31; First posted 2020-05-20 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the topic of lung cancer screening following treatment for Hodgkin lymphoma from the perspective of survivors

DETAILED DESCRIPTION:
Explore survivors' attitudes towards lung cancer and lung cancer screening Explore survivors' understanding of cancer screening as a concept and the benefits of screening and early detection Explore survivors' level of awareness of and attitudes towards their lung cancer risk Explore survivors' views on the barriers and motivating factors that would impact their decision to attend a lung cancer screening test

ELIGIBILITY:
Inclusion Criteria:

* Details held in the ADAPT database at The Christie NHS Foundation trust
* Responded to most recent ADAPT study questionnaire (April - August 2019)
* Aged 18-80
* Previously treated for Hodgkin lymphoma without evidence of relapse for at least 5 years
* Able to provide informed consent
* Treated with radiotherapy (with lung tissue in the radiotherapy field) and/or alkylating agent containing chemotherapy.

Exclusion Criteria:

* Previous or current diagnosis of lung cancer
* Stated within 2019 health questionnaire that they did not wish to be contacted
* Have participated in lung cancer screening through the Manchester Lung Health Checks

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants who have previously been treated for Hodgkin lymphoma without evidence of relapse for at least 5 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Explore survivors' attitudes towards lung cancer and lung cancer screening | 6 months
  Semi-structured interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
It is not intended to share IPD with other researchers outside the study team